CLINICAL TRIAL: NCT01299909
Title: Study Two for Development of Novel Behavioral Intervention Mindfulness Training for Smokers
Brief Title: Study Two on the Effectiveness of Mindfulness Training for Smokers
Acronym: MTS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0087; 1K23DA022471-01A1 (NIH)
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Nicotine Dependence
Keywords: Mindfulness Training for Smokers; Smoking; Smoking cessation; Addiction; behavioral intervention; Nicotine; Tobacco; Mindfulness; Meditation; MBSR; Mindfulness Based Stress Reduction; Mindfulness Based Cognitive Therapy; MBCT; Mindfulness Based Relapse Prevention; MBRP; Mindfulness Training; Nicotine Patch; Quit Line; Phone counseling; Freedom from Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation; Behavior, Addictive | interventions — Control Groups; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mindfulness Training for Smokers (Active Comparator): MTS participants will receive 8 classes of training in mindfulness meditation, access to the MTS website, and 2 weeks of nicotine patches.
  Interventions: Behavioral: Mindfulness Training for Smokers
- Integrated Training for Smokers (Active Comparator): ITS participants will receive 8 classes of training in smoking cessation strategies, access to the Freedom From Smoking online program, and 2 weeks of nicotine patches.
  Interventions: Behavioral: Integrated Training for Smokers
- Quitline (Other): Quitline participants will consist of participants who elect not to participate in the high-intensity treatments (Mindfulness Training for Smokers; Integrated Training for Smokers. This Quitline group is a Non-Randomized, Treatment as Usual group.
  Interventions: Behavioral: Quitline

INTERVENTIONS:
Behavioral: Integrated Training for Smokers — 8 classes in smoking cessation strategies, 2 weeks of nicotine patches, and access to the Freedom From Smoking online program
  Other Names: Control Group; ITS
  Arms: Integrated Training for Smokers
Behavioral: Mindfulness Training for Smokers — 8 classes of training in mindfulness meditation, 2 weeks of nicotine patches, and access to the MTS website.
  Other Names: Study Group; MTS
  Arms: Mindfulness Training for Smokers
Behavioral: Quitline — Telephone-based smoking cessation treatment via the Wisconsin Tobacco Quit Line (WTQL) consisting of 2 weeks of nicotine patches, self-help materials, an interactive website, and unlimited follow-up calls to the WTQL at no cost.
  Other Names: Non-Randomized, Treatment as Usual
  Arms: Quitline

SUMMARY:
The MTS2 study enrollment goal is N=240 adult smokers randomized to study treatments. The study design includes two randomized arms to compare matched intensive interventions and a third non-randomized option for participants who prefer not to enter an intensive intervention. It is expected that roughly 50% (120) will choose to be in the randomized intensive interventions and 50% (120) will choose to be in the non-intensive intervention. Participants who choose to be in an intensive intervention will be randomized to either Mindfulness Training for Smokers(MTS) (n = 60) or Integrated Training for Smokers (ITS)(n=60). Both MTS and ITS are smoking cessation interventions that provide 8 classes over a 6-week period and 2 weeks of nicotine patches. MTS provides and training in mindfulness whereas ITS provides training in quit smoking strategies and access to the Freedom From Smoking Online Premium Program. Participants who choose to be in a non-intensive intervention (estimated from prior recruitment data at n=120) will receive a phone-based intervention through the Wisconsin Tobacco Quit Line and 2 weeks of nicotine patches.

DETAILED DESCRIPTION:
The MTS2 Study is funded for through a five-year K23 NIH training grant (appendix) awarded to Dr. James Davis, the Principal Investigator on this protocol. The study enrollment goal is N=240 adult smokers randomized to study treatments. Based on prior recruitment numbers, it is expected that roughly 50% (120) will choose to be in an intensive intervention and 50% (120) will choose to be in the non-intensive intervention. Participants who choose to be in an intensive intervention will be randomized to either MTS (n = 60) or ITS (n=60). MTS is a smoking cessation intervention that provides 8 mindfulness classes over a 6-week period. ITS will provide participants will access to the Freedom From Smoking Online Premium Program (at no cost) plus 8 smoking cessation classes over a 6-week period. Participants who choose to be in a non-intensive intervention (n=120) will receive a phone-based intervention through the Wisconsin Tobacco Quit Line. At the Orientation Meeting, participants who decide to enter the study will be allowed to choose whether they enter an intensive or the non-intensive intervention. Intensive intervention participants will attend an additional meeting called the Introductory Meeting where they are will undergo randomization into either the MTS or ITS. The Introductory Meeting will also provide instruction on the use of nicotine patches, smoking calendars and provide intervention materials. The study employs 3 study assessment visits. Study Visit 1 follows the Orientation Meeting, Study Visit 2 is 4-weeks post-quit, Study Visit 3 is 24-weeks post-quit. All participants will receive 2 weeks of free nicotine patches and $30 for attending each of the two post-quit study visits.

The total time for the study including recruitment, intervention and participant follow-up for N = 240 will be three years. The study will recruit subjects from the Dane county region through the University of Wisconsin School of Medicine and Public Health Center for Tobacco Research and Intervention (UW-CRTI). Recruitment will take place through flyers, television, newspaper and radio advertisements.

The principal hypothesis for the study is that MTS compared to ITS will show significantly higher point prevalent Carbon Monoxide confirmed smoking abstinence rates at 4 and 24 weeks post quit. Secondary hypotheses is that study group compared to controls will show significant differences in questionnaire results that test distress, depression, anxiety, attentional control, mindfulness and quality of life and bio-physiological markers such as weight, breath holding and hair cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or over;
* Participants must express "high" motivation to quit smoking
* Participants must express willingness to attend "all" meetings for 2 months
* Smoke 5 or more cigarettes per day

Exclusion Criteria:

* Self report of alcohol use of 4 drinks or more a night on 4 or more nights per week.
* Self report of using chewing tobacco, snuff or cigars in the last week.
* High score on Patient Health Questionnaire Depression Screening Tool for severe depression and suicidal intention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Davis, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after June 2014 from Principal Investigator James Davis, MD, who is now at Duke University (james.m.davis@duke.edu).
Time Frame: Data will be available after June 2014 from Principal Investigator James Davis, MD, who is now at Duke University (james.m.davis@duke.edu).
Access Criteria: Other researchers will need to contact the Principal Investigator James Davis, MD, who is now at Duke University (james.m.davis@duke.edu).

REFERENCES:
- [Result] Davis JM, Manley AR, Goldberg SB, Smith SS, Jorenby DE. Randomized trial comparing mindfulness training for smokers to a matched control. J Subst Abuse Treat. 2014 Sep;47(3):213-21. doi: 10.1016/j.jsat.2014.04.005. Epub 2014 May 2. PMID 24957302
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700

RESULTS

PARTICIPANT FLOW:
Groups:
- Quitline: Non-Randomized, Treatment as Usual condition; participants self-selected to this group and received smoking cessation treatment via the Wisconsin Tobacco Quit Line (WTQL).
Period: Overall Study
Arm/Group | Mindfulness Training for Smokers | Integrated Training for Smokers | Quitline
Started | 68 | 67 | 40
Completed | 46 | 49 | 23
Not Completed | 22 | 18 | 17
Not completed — Lost to Follow-up | 22 | 18 | 17

BASELINE CHARACTERISTICS:
Population: This is based on enrollment - it was the number randomized. The Quitline group was a non-randomized, treatment as usual group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Training for Smokers | Integrated Training for Smokers | Quitline | Total
Number analyzed (Participants) | 68 | 67 | 40 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 67 | 40 | 175
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.24 (12.05) | 45.78 (13.35) | 45.33 (11.89) | 44.69 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 21 | 84
  Male | 39 | 33 | 19 | 91
Region of Enrollment [Number; unit: participants]
  United States | 68 | 67 | 40 | 135

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: Self-reported 7-day point-prevalence smoking abstinence (i.e., no smoking in the past 7 days) biochemically confirmed by carbon monoxide breath testing in MTS vs ITS subjects at 24 weeks post quit day.
Time Frame: 24 weeks post quit day
Population: analysis was conducted on all randomized participants
Measure: Number; unit: participants
Arm/Group | Mindfulness Training for Smokers | Integrated Training for Smokers
Number analyzed (Participants) | 68 | 67
participants | 17 | 12
Statistical Analysis 1: Comparison: Mindfulness Training for Smokers vs Integrated Training for Smokers; Test type: Superiority or Other; p = 0.35, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.67 to 3.51]

2. Secondary Outcome: Five Facet Mindfulness Questionnaire (FFMQ)
Description: The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item self-report questionnaire that assesses various components of mindfulness. Each item is rated on a 1 to 5 scale with 1=never or very rarely true and 5=very often or always true; responses are summed and then divided by 39 (the number of items). Higher scores on the FFMQ reflects a higher level of mindfulness (a better outcome).
  More information on the FFMQ is available in the following two articles:
  Baer, R. A., Smith, G. T., Hopkins, J., Krietemeyer, J., & Toney, L. (2006). Using self-report assessment methods to explore facets of mindfulness. Assessment, 13(1), 27-45, http://dx.doi.org/10.1177/1073191105283504.
  Baer,R. A., Smith,G. T., Lykins, E., Button,D., Krietemeyer, J., Sauer, S., et al. (2008). Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment, 15(3), 329-342, http://dx.doi.org/10.1177/1073191107313003.
Time Frame: 24 weeks post-quit
Population: Data are derived only from participants who completed all three study assessment visits
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Training for Smokers | Integrated Training for Smokers
Number analyzed (Participants) | 29 | 30
units on a scale | 3.72 (0.56) | 3.43 (0.48)
Statistical Analysis 1: Comparison: Mindfulness Training for Smokers vs Integrated Training for Smokers; Test type: Superiority; p = 0.03, ANOVA; df=(1,57); Mean Difference (Final Values) = 4.81

3. Secondary Outcome: Acceptance and Action Questionnaire (AAQ)
Description: The Acceptance and Action Questionnaire (AAQ) is a 9-item self-report measure of experiential avoidance. Each item is rated on a 1 to 7 scale with 1=Never true and 7=Always true; responses are summed and then divided by 9 (the number of items). The minimum score is 1 and the maximum score is 7. Higher scores equal greater levels of experiential avoidance or psychological inflexibility (a worse outcome).
  More information on the AAQ can be found in the following two articles:
  Hayes, S. C., Strosahl, K., Wilson, K. G., Bissett, R. T., Pistorello, J., Toarmino, D., et al. (2004). Measuring experiential avoidance: A preliminary test of a working model. The Psychological Record, 54(4), 553-578.
  Boelen, P. A., & Reijntjes, A. (2008). Measuring experiential avoidance: Reliability and validity of the Dutch 9-item Acceptance and Action Questionnaire (AAQ). Journal of Psychopathology and Behavioral Assessment, 30, 241-251.
Time Frame: 24 weeks post-quit
Population: Data are derived only from participants who completed all three study assessment visits
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Training for Smokers | Integrated Training for Smokers
Number analyzed (Participants) | 29 | 30
units on a scale | 3.06 (0.74) | 3.57 (0.83)
Statistical Analysis 1: Comparison: Mindfulness Training for Smokers vs Integrated Training for Smokers; Test type: Superiority; p = 0.02, ANOVA; df=(1,57); Mean Difference (Final Values) = 6.09

4. Secondary Outcome: Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale (PSS) is a self-report measure of perceived stress; the version used is a 10-item version. Each item is rated on a 0 to 4 scale with 0=Never and 4=Very Often. The minimum score is 0 and the maximum score is 40. Higher scores on the PSS reflect higher levels of perceived stress (a worse outcome).
  More information on the PSS can be found in the following article:
  Leung, D. Y., Lam, T. H., & Chan, S. S. (2010). Three versions of Perceived Stress Scale: Validation in a sample of Chinese cardiac patients who smoke. BMC Public Health, 10, 513-519
Time Frame: 24 weeks post-quit
Population: Data are derived only from participants who completed all three study assessment visits
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Training for Smokers | Integrated Training for Smokers
Number analyzed (Participants) | 29 | 30
units on a scale | 13.00 (6.48) | 16.93 (7.07)
Statistical Analysis 1: Comparison: Mindfulness Training for Smokers vs Integrated Training for Smokers; Test type: Superiority; p = 0.03, ANOVA; df=(1,57); Mean Difference (Final Values) = 4.96

ADVERSE EVENTS:
Arm/Group | Mindfulness Training for Smokers | Integrated Training for Smokers | Quitline
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67 | 0/40
Other Adverse Events (participants affected / at risk) | 0/68 | 0/67 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No